CLINICAL TRIAL: NCT00381082
Title: A Randomised, Controlled and Blinded Assessment Study of the Efficacy of MOOV Head Lice Treatment (Ego Pharmaceutical Pty. Ltd.) in the Treatment of Head Lice in Primary School Children.
Brief Title: A Randomised, Assessor-Blind, Comparative Efficacy Clinical Trial of 3 Pediculicides.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Uniquest Pty Ltd (Other)
Collaborators: Ego Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MOOV-1 Version 1 22 Sep 2004
Record Dates: First submitted 2006-09-26; First posted 2006-09-27 (Estimated); Last update posted 2006-12-12 (Estimated); Status verified 2006-12

CONDITIONS: Pediculosis
Keywords: Pediculus; capitis; lice
MeSH Terms: conditions — Lice Infestations

INTERVENTIONS:
Drug: 1) MOOV Head Lice Treatment (Ego Pharmaceutical).
Drug: Banlice Mousse Aerosol (Pfizer, Australia)
Drug: 3) KP24 Medicated Foam (Nelson Laboratories)

SUMMARY:
Objective

To compare the cure rates (defined as the complete absence of live lice, adults or nymphs, as diagnosed by wet-combing of three Australian approved head lice products for the treatment of primary school children with head lice infestation. The study design will be randomised and assessor-blind using three comparative parallel treatment groups.

The study population will consist of Queensland state primary school children (up to Year 7) with live head lice (adults or nymphs) on the hair or scalp who have not used any head lice product in the four weeks prior to the study.

DETAILED DESCRIPTION:
All products were used according to the manufacturer's instructions. KP24 and Banlice were applied twice separated by a one week interval. MOOV Head Lice Treatment was applied on Day 0, Day 7 and Day 14. The cure rate (absence of live lice) one day after the first administration for all products was a secondary outcome measure. The cure rate at 7 days after the final administration (Day 14 for Banlice or KP24 and at Day 21 for MOOV Head Lice Treatment) was the primary outcome measure. Siblings were treated if these were found to be infected as an enrolment criteria.

ELIGIBILITY:
Inclusion Criteria:

* Male or female primary school children.
* Presence of live head lice (adults or nymphs) on the hair or scalp. The presence of live lice will be determined from a visual inspection of the hair and scalp and Dry-combing of the hair. Combing will stop immediately once live lice are observed. The presence of lice eggs alone is not a sufficient condition for inclusion in the trial.
* Be available for the duration of the trial.
* Parent / Guardian is willing not to use other head lice products or methods (e.g. combs) to treat their child's head lice for 21 days after the first treatment.
* Parent / Guardian has given written informed consent to their child's participation in the trial.

Exclusion Criteria:

* History of allergies or adverse reactions to head lice products or the components of the specific products being tested.
* Treatment with any head lice product in the month prior to Day 0.
* Presence of scalp disease(s).
* If a subject has a sibling in Grade 1-7 this sibling must also be enrolled in the study and treated on Day 0 otherwise the subject must be considered ineligible for enrolment.
* Subjects must have one fixed place of residence

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 152
Dates: Start 2004-09; Study Completion 2004-11

PRIMARY OUTCOMES:
Absence of live head lice one week after the last treatment for each product (ie at Day 14 for KP24 and Banlice and at Day 21 for MOOV Head Lice Treatment)

SECONDARY OUTCOMES:
Absence of live head lice one day after the first treatment of each product

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Barker, PhD, Principal Investigator — The University of Queensland
Locations (1):
- University of Queensland, Brisbane, Queensland, Australia